CLINICAL TRIAL: NCT03554642
Title: Walkbot Robotic Training for Improvement in Gait in Sub-Acute Stroke
Brief Title: Walkbot Robotic Training for Improvement in Gait
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Burke Medical Research Institute (Other)
Collaborators: P&S Mechanics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRC532
Record Dates: First submitted 2018-05-15; First posted 2018-06-13 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Ischemic Stroke; Gait, Hemiplegic
MeSH Terms: conditions — Ischemic Stroke; Gait Disorders, Neurologic | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Sequential randomization into one of two groups within first week after admission.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Walkbot Training (Experimental): This group will receive usual inpatient care that includes at least one 60-minute session of physical therapy and an additional 30-minute session of Walkbot with Augmented Reality 5-days per week during the duration of their stay (14 days).
  Interventions: Device: Walkbot
- Physical Therapy (Active Comparator): This group will receive usual inpatient care including at least one 60-minute session of physical therapy per day, and an additional 30-minute session of standard physical therapy focused on pre-gait and/or gait training activities 5-days per week during the duration of their stay (14 days).
  Interventions: Behavioral: Physical Therapy
- Usual Care Physical Therapy (No Intervention): Participants in this group will receive usual inpatient care including at least one 60-minute session of physical therapy per day.

INTERVENTIONS:
Device: Walkbot — Walkbot is a Robot Assisted Gait Training System. This system is designed to maximize muscle strength, range of joint motion, and gait function while participants engage in a virtual reality game.
  Arms: Walkbot Training
Behavioral: Physical Therapy — 30-minute session of standard physical therapy focused on pre-gait and/or gait training activities 5-days per week during the duration of their stay (14 days).
  Arms: Physical Therapy

SUMMARY:
This clinical study will involve up to 30 ischemic stroke inpatients during their stay at Burke Rehabilitation Hospital. Participants will be randomized to receive 30 additional minutes of therapy every day, for a total of 2 weeks (14 days). One group will receive 30 minutes of standard physical therapy focused on pre-gait or gait training activities, while the experimental group will receive 30 minutes of Walkbot with Augmented Reality. Both groups will receive the same time in therapy aimed at gait training.

DETAILED DESCRIPTION:
This controlled clinical study will involve 30 ischemic stroke inpatients during their stay at Burke Rehabilitation Hospital (typical inpatient arrives 7 days post-stroke and is admitted for ~16 days).

Stroke inpatients will be sequentially randomized into one of two groups within the first week after admission. Both Groups will receive 30 additional minutes of therapy every day, for a total of 2 weeks (14 days). Group A will enroll 15 patients who will receive usual inpatient care including at least one 60-minute session of physical therapy per day, and an additional 30-minute session of standard physical therapy focused on pre-gait and/or gait training activities 5-days per week during the duration of their stay (14 days). Group B will enroll 15 patients who receive usual inpatient care that includes at least one 60-minute session of physical therapy and an additional 30-minute session of Walkbot with Augmented Reality 5-days per week during the duration of their stay (14 days). Both groups will receive the same time in therapy aimed at gait training. The extra therapy group will not exceed more than 15 minutes of pregait training before starting to walk the patient, and will spend at least 15 minutes doing active gait training per session. Patients in the treatment group will receive 30 minutes of total training on the Walkbot, excluding setup time. Primary and secondary outcomes will be collected, prior to the first therapy session. Follow up outcome measures will be collected within two days after the final interventional (study) therapy session. The amount of therapists needed for each session will be logged for every patient after Walkbot training or extra physical therapy. Borg rating of perceived exertion will be taken after each session from the patients, and NASA Task Load Index will be completed by the therapists (ie therapist load). Outcomes will be analyzed for significant differences.

ELIGIBILITY:
Inclusion Criteria:

* Cortical/subcortical ischemic stroke
* 1st time clinical stroke presentation, or prior stroke with no residual deficits affecting ambulation
* Ability to follow 2 step commands
* Fugl Meyer Sensory Score > 2
* Suitability for gait training as assessed clinically (ability to ambulate at least one step with a device/assistance)
* Height 132 cm- 200 cm; hip-knee joint length: 33 cm- 48 cm; knee joint-foot: 33 cm-48 cm

Exclusion Criteria:

* Cerebellar/brainstem stroke
* Body weight >135 kg
* Uncontrolled high blood pressure (stage 2) higher than 160 (systolic)/ 100 (diastolic)
* Cardiopulmonary system impairments affecting the ambulation test.
* Integumentary impairment: skin breakdown and bedsore around the loading area of the suspension belt
* No previous robotic intervention for ambulation training
* Significant and persistent mental illness.
* A fixed contracture or deformity in lower extremity.
* Bone instability (non-consolidated fractures, unstable spinal column, severe osteoporosis necessitating treatment with bisphosphonates).
* Other neurodegenerative disorders (Amyotrophic lateral sclerosis, Parkinsonian disorder).
* Modified Ashworth scale >3 in affected leg.
* Significant back or leg pain that creates an inability to tolerate movement.
* Decreased sensation that will impair patient's ability to percept whether the device is properly fitted
* Aphasia of a degree that would prevent the patient from communicating discomfort.
* Inability to tolerate the Walkbot device or ambulation therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer Assessment | Discharge evaluation (within 2 days after last session)
  Lower extremity impairment measure

SECONDARY OUTCOMES:
NIH Stroke Scale | Baseline assessment and discharge evaluation within 2 days after last session
  Quantitative measure of stroke-related neurological deficit; The scale is comprised of 11 items with a maximal score of 42 and minimum of 0. Higher scores indicate severe stroke.
Modified Ashworth Scale | Baseline assessment and discharge evaluation within 2 days after last session
  Measure of spasticity; Each muscle assessed is scored between 0-4, with 4 indicating rigid limbs or very severely affected.
Functional Ambulation Classification | Baseline assessment and discharge evaluation within 2 days after last session
  Clinical measure of mobility
6 Minute Walk Test | Baseline assessment and discharge evaluation within 2 days after last session
  Measures the distance that a patient can walk on a flat, hard surface in a period of 6 minutes.
10 Meter Walk Test | Baseline assessment and discharge evaluation within 2 days after last session
  Examines gait speed
Timed Up and Go | Baseline assessment and discharge evaluation within 2 days after last session
  Assesses mobility in both static and dynamic balance
Berg Balance Scale | Baseline assessment and discharge evaluation within 2 days after last session
  Assesses balance during a series of 14 tasks; higher scores indicate greater independence.
Burke Lateropulsion Scale | Baseline assessment and discharge evaluation within 2 days after last session
  5 item scale measures lateropulsion or "Pusher Syndrome" by assessing reaction to change in postural position; 0 = no lateropulsion, 17= maximum score.
Beck Depression Inventory | Baseline assessment and discharge evaluation within 2 days after last session
  21 question, multiple choice, self-report inventory to assess depression; score of 0= minimal depression, 63= severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Friel, PhD, Principal Investigator — Burke Medical Research Institute
Locations (1):
- Burke Medical Research Institute, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data with other researchers at this time.

REFERENCES:
- [Derived] Park C, Oh-Park M, Bialek A, Friel K, Edwards D, You JSH. Abnormal synergistic gait mitigation in acute stroke using an innovative ankle-knee-hip interlimb humanoid robot: a preliminary randomized controlled trial. Sci Rep. 2021 Nov 24;11(1):22823. doi: 10.1038/s41598-021-01959-z. PMID 34819515